| Role of Mirtazapin | e in / | Ameliorating | Sleep | <b>Disordered</b> | <b>Breathing</b> |
|---|---|---|---|---|---|

NCT04799782 Abdulghani Sankari, MD, PhD 4/14/2021 <u>Protocol:</u> Each subject will be studied on two separate occasions: (1) Mirtazapine vs. placebo for one week; the patients will be blinded to what medication they will be taking. The initial dose of Mirtazapine is 15 mg 30minutes before bed-time. After the one week treatment a noninvasive nasal mechanical ventilation study will be repeated to determine the hypocapnic apneic threshold. (2) Cross over medication for one week will be followed by a second noninvasive nasal mechanical ventilation study and PSG to determine the hypocapnic apneic threshold followed by two weeks washout. To assess the clinical effect of the drug on breathing during sleep a qualitative polysomnography will be performed for 2 hours the same night after taking the drug/placebo. This will allow the determination of ventilatory changes, calculation of upper airway resistance and the determination of the number of respiratory events (apnea/hypopnea index).